CLINICAL TRIAL: NCT04293380
Title: Amniotic Fluid Ischemia Modified Albumin as a Novel e Prenatal Diagnostic Marker for Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Guven, professor, Karadeniz Technical University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: suleymanG
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Down Syndrome; Prenatal Stress; Cytokines
Keywords: Down Syndrome; Prenatally; ischemic modified album; cytokines; amniyosyntesis
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal karyotype (Other): During the prenatal evaluation, IMA and cytokine values in amniotic fluid will be compared in cases with down syndrome and normal karyotype.
  Interventions: Procedure: amniosyntesis
- down syndrome (Other): During the prenatal evaluation, IMA and cytokine values in amniotic fluid will be compared in cases with down syndrome and normal karyotype.
  Interventions: Procedure: amniosyntesis

INTERVENTIONS:
Procedure: amniosyntesis

SUMMARY:
Down syndrome is the most common genetic disorder in the society that causes mental retardation. Today, screening tests (combined test, triple screening, ultrasonography and age) are performed for the diagnosis of down syndrome for all pregnant women. As a result of screening tests, amniocentesis is performed as a diagnostic test for the group at risk. Chromosome analysis from amniotic fluid requires a 3-week period for chromosome cultures to yield results. Several levels of biochemical markers, such as organic acids and pyridoxine metabolites, have been found to be elevated in the amniotic fluid. The investigators also plan to investigate ischemia-modified albumin, hepatocyte growth factor level in amniotic fluid.

DETAILED DESCRIPTION:
The alpha feto protein level showing liver function is lower in babies with Down syndrome and this biochemical marker is one of the basic parameters of triple screening.

If these babies have insufficient liver function, then it is likely that there is a decrease in hepatocyte growth factor in these babies. Free E3 is higher in Down syndrome than normal pregnant women. Placental hyperfunction, fetal hypofunction (especially based on fetal liver) is accepted as the hypothetical cause of these two conditions in Down syndrome. In this study, the investigators think that the real cause of this condition is secondary to fetal partial hypoxia. For this purpose, the investigators plan to look at the level of IMA in amniotic fluid. However, Güven et al. In his study, an increased rate of ischemia-modified albumin was found in the amnion levels of mothers who had high triple screening tests but had no down syndrome in their babies. In this study, it is aimed to find a change in amniotic fluid that can help in the diagnosis of down syndrome. In our opinion, in cases of down syndrome, there will be an increase in IMA in the amniotic fluid secondary to ischemia, which is more severe than the false triple test positivity.

In our university, chromosome analyzes are made from amnion fluids sent to the Duzen laboratory. This laboratory hides amniotic fluid of patients with down syndrome (in the context of an agreement between our university and the laboratory). Within the scope of the research, amniotic fluids of 20 cases diagnosed with down syndrome in the Department of Obstetrics and Gynecology of KTU Faculty of Medicine will be obtained from the regulation laboratory and necessary biochemical evaluations will be performed. As the control group, amniotic fluids will be provided by 60 patients with normal amniocentesis results. The demographic factor, obstetric history and gynecological history information of all cases will be recorded in the questionnaire prepared by one of the researchers. 2 cc amnion sample of the patients with Down syndrome diagnosis and control group will be taken into the biochemistry tube and serum IMA and HGF values will be measured in KTU Faculty of Medicine, Department of Biochemistry. As a result, amnion IMA, HGF values of 20 cases diagnosed with down syndrome and amnion IMA, HGF values of 60 cases with down syndrome will be entered into SPSS 10.5 for Windows environment and their mean values will be compared.

According to the results, amniotic fluid IMA values of the study group and control group will be compared. Thus, it is aimed to eliminate the burden that the chromosome culture will bring to the national economy with an evaluation made in a routine laboratory in cases diagnosed with down syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 20 cases diagnosed with down syndrome in the Duzen laboratory chromosome culture
* 74 cases which are normal in the Duzen laboratory chromosome culture

Exclusion Criteria:

- absent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — on pregnant women
Enrollment: 94 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
The IMA levels | immediately after the procedure
  The IMA levels in our study group was higher than control group.

CONTACTS AND LOCATIONS:
Overall Officials: suleyman guven, professor, Principal Investigator — karadeniz thecnical universty; erhan huseyın comert, Study Chair — gole goverment hospital; emine seda guvendag guven, Study Chair — karadeniz thecnical universty
Locations (1):
- Karadeniz Technical Universty Medical School, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No